CLINICAL TRIAL: NCT01668940
Title: Effectiveness of a Natural Non-medicinal Freezie Remedy to Alleviate Morning Sickness
Brief Title: Freezie Remedy to Alleviate Morning Sickness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study PI left the institution in early 2015.
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Shinya Ito, Division Head, Clinical Pharmacology and Toxicology, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000031589
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Morning Sickness
Keywords: Morning Sickness; Lillipops Iced Soothies; Pregnancy; Obstetrics
MeSH Terms: conditions — Morning Sickness

STUDY DESIGN:
Intervention Model Description: Four parallel groups: 1) Lillipops Group (4 flavours): 2) Ginger Lillipops Group; 3) Mr. Freeze Control Group; 4) Natural Course Group. The main comparison is Group 1 vs Group 3.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A computerized randomization table will be prepared by a third party who is not otherwise involved in the study. After a participant has given consent to enrol in the study, the next participant number in sequence will be assigned and the appropriate corresponding sealed envelope will be opened by the study coordinator, determining which product (if any) the participant will receive. The boxes will be given unique codes depending on whether they contain Lillipops (4 flavours), Ginger Lillipops or Mr. Freeze freezies, and the different flavours will also be coded. Participants will be shown a list of the ingredients that are found in Lillipops and Mr. Freeze freezies to ensure that they do not have allergies or take medications that interact with any ingredient(s) that they may be asked to consume.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lillipops Iced Soothies (4 flavours) (Experimental): Initially, women will be given 1 multiflavour box of Lillipop samples minus the ginger flavour (4 flavours). Each box contains 24 freezies (20 mL each), 6 of each flavor. They will be told to eat the freezies as needed to alleviate symptoms, up to a maximum of 12 per day, and to not have any other popsicles, freezies or any ginger products throughout the duration of the study (7 days). They can request an additional multiflavour box of freezies at each follow-up, as needed.
  All participants will initially receive counselling and advice by the Motherisk NVP Counsellor about symptom management. This includes advice about dietary, non-medicinal and medical treatments as per the Motherisk NVP protocol
  Interventions: Other: Lillipops Iced Soothies (4 flavours)
- Lillipop Iced Soothies (Ginger flavour) (Experimental): Initially, women will be given 1 Ginger flavor box of Lillipop samples. Each box contains 24 freezies (20 mL each). Each 20ml contains 80mg of dried ginger root. They will be told to eat the freezies as needed to alleviate symptoms, up to a maximum of 12 a day and to not have any other popsicles, freezies or other ginger products throughout the duration of the study (7 days). Due ginger's antiemetic property, a maximum daily dose is up to 1000mg/day of dried ginger root powder in pregnancy.They can request an additional box of freezies at each follow-up, as needed.All participants will initially receive counselling and advice by the Motherisk NVP Counsellor about symptom management. This includes advice about dietary, non-medicinal and medical treatments as per the Motherisk NVP protocol.
  Interventions: Other: Lillipop Iced Soothies (Ginger flavour)
- Mr. Freeze Freezies (4 flavours) (Active Comparator): Initially, women will be given 1 multiflavour box of Mr. Freeze samples. Each box contains 24 freezies (20 mL each), 6 of each flavor. They will be told to eat the freezies as needed to alleviate symptoms, up to a maximum of 12 per day, and to not have any other popsicles, freezies or any ginger products throughout the duration of the study (7 days). They can request an additional multiflavour box of freezies at each follow-up, as needed.
  All participants will initially receive counselling and advice by the Motherisk NVP Counsellor about symptom management. This includes advice about dietary, non-medicinal and medical treatments as per the Motherisk NVP protocol
  Interventions: Other: Mr. Freeze Freezies
- Natural Course Group (No Intervention): Women will not receive any freezies and will be asked to not have any other popsicles, freezies or any ginger products throughout the duration of the study (7 days).
  All participants will initially receive counselling and advice by the Motherisk NVP Counsellor about symptom management. This includes advice about dietary, non-medicinal and medical treatments as per the Motherisk NVP protocol

INTERVENTIONS:
Other: Lillipops Iced Soothies (4 flavours) — Lillipops Iced Soothies are naturally flavoured freezies developed in the United Kingdom for women with morning sickness. They are available in 5 different flavours: grapefruit and tangerine, lemon and mint, chamomile and orange, lime and vanilla, and ginger. The flavours are derived from steam distillation of the peels (grapefruit, tangerine, lemon, orange, lime), mint leaves, and chamomile flowers to release and collect their essential oils. Vanilla pods and ginger are macerated and their resin is used. These flavours were chosen because they may provide relief of symptoms as they are either traditional remedies for NVP, such as ginger, or soothing and refreshing flavours, such as chamomile, vanilla and citrus.
  Arms: Lillipops Iced Soothies (4 flavours)
Other: Mr. Freeze Freezies — There are other commercially available freezies, such as Mr. Freeze. Mr. Freeze freezies contain simulated flavours of watermelon, cherry, blue raspberry and cream soda. However, there have been no reports, studies or claims that they are effective as a remedy for the treatment of NVP.
  Arms: Mr. Freeze Freezies (4 flavours)
Other: Lillipop Iced Soothies (Ginger flavour) — Lillipops Iced Soothies are naturally flavoured freezies developed in the United Kingdom for women with morning sickness. They are available in 5 different flavours: grapefruit and tangerine, lemon and mint, chamomile and orange, lime and vanilla, and ginger.The flavours are derived from steam distillation of the peels (grapefruit, tangerine, lemon, orange, lime), mint leaves, and chamomile flowers to release and collect their essential oils. Vanilla pods and ginger are macerated and their resin is used. These flavours were chosen because they may provide relief of symptoms as they are either traditional remedies for NVP, such as ginger, or soothing and refreshing flavours, such as chamomile, vanilla and citrus.
  Arms: Lillipop Iced Soothies (Ginger flavour)

SUMMARY:
The primary objective of this study is to assess the effectiveness of Lillipops in the improvement of morning sickness symptoms. Secondary objectives are to assess if there are any changes to concurrent symptoms that may intensify NVP, such as metallic taste or gastrointestinal issues (e.g. heartburn, acid reflux, indigestion and gas), as well as preference for freezie flavours.

DETAILED DESCRIPTION:
Nausea and vomiting of pregnancy (NVP) is the most common medical condition of pregnancy, also known as morning sickness which affects up to 80% of pregnant women. Lillipops Iced Soothies are naturally flavoured freezies developed in the United Kingdom for women with morning sickness. They are available in 5 different flavours: grapefruit and tangerine, lemon and mint, chamomile and orange, lime and vanilla, and ginger. The flavours are derived from steam distillation of the peels (grapefruit, tangerine, lemon, orange, lime), mint leaves, and chamomile flowers to release and collect their essential oils. Vanilla pods and ginger are macerated and their resin is used. These flavours are chosen because they may provide relief of symptoms as they are either traditional remedies for NVP, such as ginger, or soothing and refreshing flavours, such as chamomile, vanilla and citrus.

This study hypothesizes that using Lillipops Iced Soothies will reduce the severity of NVP symptoms according to the PUQE-24 (pregnancy-unique quantification of emesis and nausea) scoring system for nausea and vomiting of pregnancy. In addition, we hypothesize concurrent symptoms that may intensify NVP, such as metallic taste or gastrointestinal disorders (e.g. heartburn, acid reflux, indigestion and gas), will be alleviated. We hypothesize that improvements to NVP and concurrent symptoms will be greater with Lillipop freezies compared to another commercially available freezie.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy between 4 and 12 weeks gestation.
* Pregnant women with NVP, regardless of treatment (if any) for their NVP.
* Provide the signed informed consent form prior to initial interview.
* Able to come in person to Sick Kids or meet at an agreed location.

Exclusion Criteria:

* Gestational age beyond 12 weeks of pregnancy.
* Pregnant women less than 18 years of age.
* Women who are not proficient in the English language.
* Unable to consume any of the ingredients listed in Lillipops or Mr. Freeze freezies due to allergies, medication interactions or other reasons.
* Women refusing to avoid sources of ginger products for the duration of the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shinya Ito, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Mr. Freeze Freezies (4 Flavours): Initially, women will be given 1 multiflavour box of Mr. Freeze samples. Each box contains 24 freezies (20 mL each), 6 of each flavor. They will be told to eat the freezies as needed to alleviate symptoms, up to a maximum of 12 per day, and to not have any other popsicles, freezies or any ginger products throughout the duration of the study (7 days). They can request an additional multiflavour box of freezies at each follow-up, as needed.
  All participants will initially receive counselling and advice by the Motherisk NVP Counsellor about symptom management. This includes advice about dietary, non-medicinal and medical treatments as per the Motherisk NVP protocol
  Mr. Freeze freezies contain simulated flavours of watermelon, cherry, blue raspberry and cream soda. However, there have been no reports, studies or claims that they are effective as a remedy for the treatment of NVP.
Period: Overall Study
Arm/Group | Lillipops Iced Soothies (4 Flavours) | Lillipop Iced Soothies (Ginger Flavour) | Mr. Freeze Freezies (4 Flavours) | Natural Course Group
Started | 17 | 14 | 9 | 14
Completed | 17 (Data collection was completed, but data analysis did not occur due to study closure.) | 14 (Data collection was completed, but data analysis did not occur due to study closure.) | 9 (Data collection was completed, but data analysis did not occur due to study closure.) | 14 (Data collection was completed, but data analysis did not occur due to study closure.)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lillipops Iced Soothies (4 Flavours) (Experimental): Initially, women will be given 1 multiflavour box of Lillipop samples minus the ginger flavour (4 flavours). Each box contains 24 freezies (20 mL each), 6 of each flavor. They will be told to eat the freezies as needed to alleviate symptoms, up to a maximum of 12 per day, and to not have any other popsicles, freezies or any ginger products throughout the duration of the study (7 days). They can request an additional multiflavour box of freezies at each follow-up, as needed.
  All participants will initially receive counselling and advice by the Motherisk NVP Counsellor about symptom management. This includes advice about dietary, non-medicinal and medical treatments as per the Motherisk NVP protocol
- Lillipop Iced Soothies (Ginger Flavour) (Experimental): Initially, women will be given 1 Ginger flavor box of Lillipop samples. Each box contains 24 freezies (20 mL each). Each 20ml contains 80mg of dried ginger root. They will be told to eat the freezies as needed to alleviate symptoms, up to a maximum of 12 a day and to not have any other popsicles, freezies or other ginger products throughout the duration of the study (7 days). Due ginger's antiemetic property, a maximum daily dose is up to 1000mg/day of dried ginger root powder in pregnancy.They can request an additional box of freezies at each follow-up, as needed.All participants will initially receive counselling and advice by the Motherisk NVP Counsellor about symptom management. This includes advice about dietary, non-medicinal and medical treatments as per the Motherisk NVP protocol.
- Mr. Freeze Freezies (4 Flavours) (Active Comparator): Initially, women will be given 1 multiflavour box of Mr. Freeze samples. Each box contains 24 freezies (20 mL each), 6 of each flavor. They will be told to eat the freezies as needed to alleviate symptoms, up to a maximum of 12 per day, and to not have any other popsicles, freezies or any ginger products throughout the duration of the study (7 days). They can request an additional multiflavour box of freezies at each follow-up, as needed.
  All participants will initially receive counselling and advice by the Motherisk NVP Counsellor about symptom management. This includes advice about dietary, non-medicinal and medical treatments as per the Motherisk NVP protocol
- Natural Course Group (No Intervention): Women will not receive any freezies and will be asked to not have any other popsicles, freezies or any ginger products throughout the duration of the study (7 days).
  All participants will initially receive counselling and advice by the Motherisk NVP Counsellor about symptom management. This includes advice about dietary, non-medicinal and medical treatments as per the Motherisk NVP protocol
- Total: Total of all reporting groups
Arm/Group | Lillipops Iced Soothies (4 Flavours) (Experimental) | Lillipop Iced Soothies (Ginger Flavour) (Experimental) | Mr. Freeze Freezies (4 Flavours) (Active Comparator) | Natural Course Group (No Intervention) | Total
Number analyzed (Participants) | 17 | 14 | 9 | 14 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 14 | 9 | 14 | 54
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 31 [25 to 37.9] | 33.9 [26.6 to 40.8] | 33.6 [27.3 to 41.5] | 31.8 [27.1 to 38.9] | 32.4 [25 to 41.5]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All participants female as per study inclusion criteria. No analysis was completed due to study termination/closure.
  Participants
    Female | 17 | 14 | 9 | 14 | 54
    Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: All participants recruited in Canada as per study inclusion criteria (i.e. ability to meet at study site or nearby location). No analysis was completed due to study termination/closure.
  participants
    Canada | 17 | 14 | 9 | 14 | 54

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Nausea and Vomiting of Pregnancy (NVP)
Description: To assess the effectiveness of Lillipops in the improvement of NVP symptoms. The primary endpoint of interest is the severity of NVP as compared between the 4 groups, defined according to the PUQE-24 (pregnancy-unique quantification of emesis and nausea) scoring system for nausea and vomiting of pregnancy that was developed and validated by Motherisk.
Time Frame: Baseline, +1, +3, +5, +7 days
Population: The study was terminated due to the original study PI's departure, and the final analyses have not been conducted. The study file has been locked in 2015 after the official study closure.
Arm/Group | Lillipops Iced Soothies (4 Flavours) | Lillipop Iced Soothies (Ginger Flavour) | Mr. Freeze Freezies (4 Flavours) | Natural Course Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Concurrent Symptoms
Description: To assess if there are any changes to concurrent symptoms that may intensify NVP, such as metallic taste or gastrointestinal issues (e.g. heartburn, acid reflux, indigestion and gas). The secondary endpoint of interest is the effect of the 4 groups on the status of concurrent symptoms that may intensify NVP, such as metallic taste or gastroesophageal reflux disease, as well as preference for freezie flavours, according to the PUQE-24 (pregnancy-unique quantification of emesis and nausea) scoring system for nausea and vomiting of pregnancy that was developed and validated by Motherisk.
Time Frame: Baseline, +1, +3, +5, +7 days
Reporting Status: Not Posted

3. Secondary Outcome: Freezie Flavour Preference
Description: To assess preference for freezie flavours.
Time Frame: Baseline, +1, +3, +5, +7 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Lillipops Iced Soothies (4 Flavours) | Lillipop Iced Soothies (Ginger Flavour) | Mr. Freeze Freezies (4 Flavours) | Natural Course Group
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/9 | 0/14
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/9 | 0/14

LIMITATIONS AND CAVEATS:
Study was terminated prior to completion. Data collected from participants was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No